CLINICAL TRIAL: NCT05910385
Title: Sexuality After Tubal Sterilization by Conventional Abdominal Laparoscopy or Vaginal Natural Orifice Transluminal Endoscopy (vNOTES) : a Randomised Controlled Trial
Brief Title: TUbal LIgation Per Differents Endoscopic Routes and Sexuality (TULIPES)
Acronym: TULIPES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RBHP 2021 CURINIER 2; 2021-A02263-38 (Other: ANSM)
Record Dates: First submitted 2023-04-25; First posted 2023-06-18 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Gynecologic Surgery
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, single-blind, two-parallel, bicentric therapeutic trial comparing two referenced surgical techniques
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic (Active Comparator)
  Interventions: Procedure: laparoscopy
- vnotes (Experimental)
  Interventions: Procedure: vnotes

INTERVENTIONS:
Procedure: laparoscopy — tubal ligation by laparoscopy or vnotes technique
  Arms: laparoscopic
Procedure: vnotes — tubal ligation by laparoscopy or vnotes technique
  Arms: vnotes

SUMMARY:
The goal of this clinical trial is compare the quality of sexual life at 6 months after tubal ligation, depending on whether it was performed by abdominal laparoscopy or by vNOTES, on the basis of a non-inferiority hypothesis. Participants will answer on the FSFI-19 questionnaire and quality of sexual life will be evaluated according to the score obtained at 6 months post-operative compared to pre-operative.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman, eligible for tubal ligation by total salpingectomy or tubal section coagulation, sexually active at the time of inclusion
* Able to give informed consent to participate in research
* Affiliated to a social security system.

Exclusion Criteria:

* Current pregnancy or breastfeeding
* Indications of another concomitant surgical procedure (other than procedure on the appendix)
* History of upper genital infection
* Proven or suspected rectovaginal endometriosis on clinical examination
* History of rectal surgery
* Virgin patient
* Any concomitant pathology deemed incompatible with the study.
* Uncured COVID or SARS-COv2 positivity dated less than 3 days prior to surgery.
* Protected adult patient, under guardianship or curatorship
* Patients not affiliated to the social security system
* Patients who do not speak French
* Patients under legal protection
* Refusal to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
quality of sexual life | 6 months
  To compare, on the basis of a non-inferiority hypothesis, the quality of sexual life at 6 months after tubal ligation, depending on whether it is performed by abdominal laparoscopy or by vNOTES, using the Female Sexual Function Index - 19 (FSFI-19) questionnaire (19 questions with 6 possible answers for each, with scores ranging from 0=worse outcome to 5=better outcome).

SECONDARY OUTCOMES:
characteristics of the course of surgery for tubal ligation (duration of installation and intervention in minutes) | 6 months
  - Compare the characteristics of the course of surgery for tubal ligation (duration of installation and intervention in minutes), depending on whether it is performed by abdominal laparoscopy or by vNOTES.
postoperative pain | 6 months
  Compare the consequences of tubal ligation, depending on whether it is performed by abdominal laparoscopy or by vNOTES, in term of postoperative pain, using EVA Scale (from 0 to 10).
consumption of peroperative analgesics. | 6 months
  Compare the consequences of tubal ligation, depending on whether it is performed by abdominal laparoscopy or by vNOTES, in term of consumption of peroperative analgesics (e.g. name of the analgesics, dose and duration of intake in days).
consumption of postoperative analgesics. | 6 months
  Compare the consequences of tubal ligation, depending on whether it is performed by abdominal laparoscopy or by vNOTES, in term of consumption of postoperative analgesics (e.g. name of the analgesics, dose and duration of intake in days).
per and post-operative complications | 6 months
  - Compare the consequences of tubal ligation, depending on whether it is performed by abdominal laparoscopy or by vNOTES, in terms of per and post-operative complications.
patient satisfaction | 6 months
  - Compare the consequences of tubal ligation, depending on whether it is performed by abdominal laparoscopy or by vNOTES, in term of patient satisfaction (Very dissatisfied, Moderately dissatisfied, Neither satisfied nor dissatisfied, Moderately satisfied, Very satisfied).
quality of life after surgery | 6 months
  - Compare the consequences of tubal ligation, depending on whether it is performed by abdominal laparoscopy or by vNOTES, in term of patient quality of life after surgery, using EQ-5D-5L questionnaire (with five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems).
number of days of sick leave | 6 months
  - Compare the number of days of sick leave, depending on whether it is performed by abdominal laparoscopy or by vNOTES.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Curinier, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CH d'Issoire, Issoire